NCT Number: NCT06375421

Title: Pilot and Feasibility of MEMI for Chronic Traumatic Brain Injury

**Document Date:** 07/16/2025

## NCT06375421 - Statistical analysis plan

For this pilot study, we calculated descriptive statistics for participant characteristics, engagement (number of sessions completed), acceptability (Acceptability of Intervention Measure), and preliminary efficacy using R. Baseline participant characteristics were calculated for each group (TBI and non-injured comparison groups). Engagement, acceptability, and preliminary efficacy analyses were conducted within each group between the two conditions (Intervention: MEMI and Active Comparator: Blocked). For preliminary efficacy, we used paired-samples t-tests within each group to compare free recall at the 1-week assessment between the two conditions. We also conducted supplementary analyses assessing cued word form recall and cued definition recall at the 1-week assessment. Analyses were conducted using a complete-case approach.